CLINICAL TRIAL: NCT00933192
Title: The Relationship Between Muscle Morphology and Muscle Strength
Status: Completed | Type: Observational
Sponsor: Karl Landsteiner Institute of Remobilization and Functional Health (Other)
Responsible Party: Karl Landsteiner Institute of Remobilization and Functional Health, Institute of Physical Medicine and Rehabilitation
Other Study IDs: muscle ultrasound
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Skeletal Muscle Ultrasound; Isometric Muscle Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group 1: young healthy patients
  Interventions: Device: Siemens Acuson Antares ultrasound
- Group 2: old healthy patients
  Interventions: Device: Siemens Acuson Antares ultrasound

INTERVENTIONS:
Device: Siemens Acuson Antares ultrasound — skeletal muscle ultrasound of the musculus quadriceps, on two different days, two observers

SUMMARY:
The evaluation of skeletal muscle strength in severly ill or cognitive impaired patients is an unresolved problem especially during the rehabilitation process. The aim of this study is to correlate morphological parameters assessed with muscle ultrasound and isometric muscle strength to establish an objective progression parameter for rehabilitation therapies.

ELIGIBILITY:
Inclusion Criteria:

* group 1: patients between 18 and 35 years
* group 2: patients between 60 and 80 years

Exclusion Criteria:

* neuromuscular diseases
* hip or knee prosthesis in the investigated leg
* any trauma of the hip, knee or ankle of the investigated leg during the last 12 months
* cognitive impairments
* pregnancy
* diabetes mellitus Type II
* acute or chronic pain in the investigated leg
* chronic maligne or non - maligne diseases (of the heart, lung or kidney)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatients or inpatients of the institute of physical medicine and rehabilitaion
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Karl Landsteiner Institute of Remobilisation and Functional Health, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Strasser EM, Draskovits T, Praschak M, Quittan M, Graf A. Association between ultrasound measurements of muscle thickness, pennation angle, echogenicity and skeletal muscle strength in the elderly. Age (Dordr). 2013 Dec;35(6):2377-88. doi: 10.1007/s11357-013-9517-z. Epub 2013 Mar 2. PMID 23456136